CLINICAL TRIAL: NCT00037167
Title: Impact of Running Poles on Older Adult Exercise Walking
Brief Title: Effects of Exercise Poles on Older Adults During Exercise Walking
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: Ball State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44AR048029 (NIH); NIAMS-071
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Movement Disorders; Aging
Keywords: Fall-Prevention; Balance; Musculoskeletal Systems; Protective Devices; Gait; Equilibrium; Accidental Falls; Frail Elderly
MeSH Terms: conditions — Movement Disorders

INTERVENTIONS:
Device: Exercise poles

SUMMARY:
This study uses a patented type of exercise poles, developed to assist runners rehabilitating from lower body injuries. These poles may offer older adults improved stability, reduced fear of falling, and lessened lower body pain when exercise walking.

DETAILED DESCRIPTION:
Phase 1 (being concluded as of Feb 2002) used 18 older adults to investigate prototype versions of the running poles. Preliminary results, after 3 months of testing, indicate the poles are safe and effective. Phase 2 will use improved versions of the poles, which are currently in development, with a group of around 125-150 subjects over a longer length of time (12 months). Changes in walking gait quality, balance, strength, body composition, exercise adherence, and subjective perceptions of wellness will be assessed before, during, and after the 12 month exercise session.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80
* Normal gait

Exclusion Criteria:

* Inability to walk continuously for 5 minutes
* Contraindication from a personal physician
* Height over 6'2" or weight over 200 lbs (due to limitations of existing pole design)
* Mild to severe cognitive impairment

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150
Dates: Start 2001-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin van Breems, Principal Investigator — Martinus Van Breems, Inc.
Locations (1):
- School of Physical Education, Biomechanics Lab, Muncie, Indiana, United States